CLINICAL TRIAL: NCT00816894
Title: D-serine Antipsychotic Monotherapy for Treatment Refractory Schizophrenia
Brief Title: D-serine Monotherapy for Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herzog Hospital (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Heresco-Levi Uriel, Princepal Investigator, Herzog Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Heresco CTIL147-08; 20080201
Record Dates: First submitted 2009-01-01; First posted 2009-01-05 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; treatment resistance; D-serine; Olanzapine; treatment refractory schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-serine arm (Experimental): 6 week fixed dose phase with D-serine 1500 mg/day to be increased starting from week two to 3000 mg/day followed by a 4 week flexible dose phase allowing for two 500 mg/day dose changes.
  Interventions: Drug: D-serine
- Olanzapine arm (Active Comparator): 6 week fixed dose phase with Olanzapine 15 mg/day to be increased starting from week two to 30 mg/day followed by a 4 week flexible dose phase allowing for two 5 mg/day dose changes.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: D-serine — 6 week fixed dose phase with D-serine 1500 mg/day to be increased starting from week two to 3000 mg/day followed by a 4 week flexible dose phase allowing for two 500 mg/day dose changes
  Other Names: DSR
  Arms: D-serine arm
Drug: Olanzapine — 6 week fixed dose phase with Olanzapine 15 mg/day to be increased starting from week two to 30 mg/day followed by a 4 week flexible dose phase allowing for two 5 mg/day dose changes.
  Other Names: Zyprexa
  Arms: Olanzapine arm

SUMMARY:
A first generation of clinical studies, performed during the last decade, demonstrates that adjuvant treatment with compounds that enhance NMDAR-mediated neurotransmission due to their agonistic activity at the NMDAR-associated glycine (GLY) site (e.g. GLY, D-serine (DSR)) leads to significant symptom reductions in chronic schizophrenia patients.Furthermore, preliminary findings suggest that treatment with NMDAR-GLY site modulators may also be beneficial as antipsychotic monotherapy In the proposed project, during a three year period, 60 schizophrenia patients that fulfill treatment resistance criteria will be randomly entered in a 10 week, two phase (fixed/flexible dose), parallel group, double blind controlled study assessing the efficacy of olanzapine (OLA) (up to 40 mg/day) vs. DSR (up to 4000 mg/day) as antipsychotic monotherapy.Clinical, neurocognitive, electrophysiological, and amino acids (i.e. GLY, DSR) levels assessments will be performed during the study. The specific aims of the proposed project are: 1) to assess the efficacy and safety of DSR as a new medication for treatment refractory schizophrenia, and 2) to assess DSR effects in terms of relevant amino acids serum levels, neurocognitive performance, and relevant brain electrophysiological parameters. The overall importance of the proposed project consists of its potential to lay the foundations for an innovative type of intervention for treatment resistant schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70;
2. Diagnosis of schizophrenia/schizoaffective disorder according to DSM-IV criteria.
3. Stable dose antipsychotic treatment for at least 4 weeks;
4. Treatment refractoriness according to Kane et al.(1988) criteria.

Exclusion Criteria:

1. Meeting criteria for other DSM-IV Axis I diagnoses ;
2. Substance abuse or alcoholism during entire lifetime;
3. Are judged clinically to be at suicidal or homicidal risk;
4. Female patients who are pregnant or lactating; female patients who are not pregnant or lactating, if sexually active, must be using medically accepted means of contraception;
5. Patients with known intolerance to OLA treatment or who have failed an adequate trial of OLA (at least 6 weeks) at high doses (20 mg/day or higher);
6. Patients treated with depot antipsychotics or ECT within the eight weeks prior to study entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
PANSS change scores. | ~ biweekly throughout the study
side effects | ~ biweekly throughout the study

SECONDARY OUTCOMES:
% treatment responders | End of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Ezrath Nashim - Herzog Memorial Hospital, Jerusalem, Israel